CLINICAL TRIAL: NCT04290143
Title: Introducing a New and Validated Placebo Development Method to Healing Water Based Rehabilitation Research
Brief Title: Placebo Development and Validation for Healing Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Collaborators: Harkány Spa Hospital, Harkány, Hungary (Unknown); National Research, Development and Innovation Office, Budapest, Hungary (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OTKA_131531_PLACEBO
Record Dates: First submitted 2020-02-17; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Balneology
Keywords: medical water; healing water; placebo

STUDY DESIGN:
Intervention Model Description: double blind study for testing a placebo development method
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both medical water and tap water will be colored. The temperature and the pH of the tap water will be adjusted to the temperature pH of the healing water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colored healing water (Active Comparator): Colored medical water in a bath tub. A single 20 minutes-long treatment will be performed.
  Interventions: Other: Colored healing water; Other: Placebo treatment (colored tap water)
- Placebo - Colored tap water (Placebo Comparator): Colored tap water. The temperature and the pH of the tap water will be adjusted to the temperature pH of the healing water. A single 20 minutes-long treatment will be performed.
  Interventions: Other: Colored healing water; Other: Placebo treatment (colored tap water)

INTERVENTIONS:
Other: Colored healing water — Patients will be treated with colored healing water for 20 minutes.
Other: Placebo treatment (colored tap water) — Patients will be treated with colored tap water for 20 minutes.

SUMMARY:
The study aimed to develop and validate an easy-to use cheap method capable of producing placebo from tap water.

DETAILED DESCRIPTION:
Introduction: The beneficial health effects of healing waters have been reported by numerous studies. However, the lack of proper placebo substance makes the "medication-like" investigation of healing waters difficult. The investigators aimed to develop and validate an easy-to use cheap method capable of producing placebo from tap water.

Methods: Both medical water and tap water will be colored. The temperature and the pH of the tap water will be adjusted to the temperature pH of the healing water. The patients will be divided into two groups, colored healing water and placebo group. A single 20 minutes-long treatment will be performed in bath tubs. Considering the healing waters odor, the treatment will be given in the same room. Patients will be asked to tell whether they are treated with colored healing water or placebo or could not tell. Questions will be asked before the treatment, 10 minutes after the beginning of the treatment, immediately after the end of the treatment and after shower. The study will be performed in a double blind setup. Patients will be scored, one point for each correct answer.

Target patient number:174

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the study
* age between 18-80 years

Exclusion Criteria:

* patients physically unable to enter or exit the bath tub
* autoimmune diseases
* any kind of malignity
* acute inflammation
* infection
* acute coronary syndrome or recent surgical interventions (6 month before enrollment)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Number of participants who responded 'placebo,' to question 1 | prior to treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded 'colored healing water' to question 1 | prior to treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded ' could not tell' to question 1 | prior to treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded 'placebo,' to question 2 | 10 minutes after the beginning of treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded 'colored healing water' to question 2 | 10 minutes after the beginning of treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded ' could not tell' to question 2 | 10 minutes after the beginning of treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded 'placebo,' to question 3 | Immediately after the end of the treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded 'colored healing water' to question 3 | Immediately after the end of the treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded ' could not tell' to question 3 | Immediately after the end of the treatment
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded 'placebo,' to question 4 | After taking a sower (within 15 minutes after the end of the treatment)
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded 'colored healing water' to question 4 | After taking a sower (within 15 minutes after the end of the treatment)
  The measurement is performed by a questionnaire filled in accordingly by an investigator
Number of participants who responded ' could not tell' to question 4 | After taking a sower (within 15 minutes after the end of the treatment)
  The measurement is performed by a questionnaire filled in accordingly by an investigator

CONTACTS AND LOCATIONS:
Overall Officials: Katalin Dr Szendi, MD, PhD, Principal Investigator — University of Pecs
Locations (2):
- Hungary (2):
  - Harkány Thermal Rehabilitation Centre, Harkány, Baranya
  - Katalin Dr Szendi, Pécs, Baranya

IPD SHARING:
Plan to Share IPD: No
Not necessary for the study purpose.

REFERENCES:
- [Background] Bender T, Balint G, Prohaszka Z, Geher P, Tefner IK. Evidence-based hydro- and balneotherapy in Hungary--a systematic review and meta-analysis. Int J Biometeorol. 2014 Apr;58(3):311-23. doi: 10.1007/s00484-013-0667-6. Epub 2013 May 16. PMID 23677421
- [Background] Szucs L, Ratko I, Lesko T, Szoor I, Genti G, Balint G. Double-blind trial on the effectiveness of the Puspokladany thermal water on arthrosis of the knee-joints. J R Soc Health. 1989 Feb;109(1):7-9. doi: 10.1177/146642408910900104. No abstract available. PMID 2494341
- [Background] Matsumoto S. Evaluation of the Role of Balneotherapy in Rehabilitation Medicine. J Nippon Med Sch. 2018;85(4):196-203. doi: 10.1272/jnms.JNMS.2018_85-30. PMID 30259887
- [Background] Morer C, Roques CF, Francon A, Forestier R, Maraver F. The role of mineral elements and other chemical compounds used in balneology: data from double-blind randomized clinical trials. Int J Biometeorol. 2017 Dec;61(12):2159-2173. doi: 10.1007/s00484-017-1421-2. Epub 2017 Aug 28. PMID 28849535
- [Background] Hanzel A, Horvat K, Molics B, Berenyi K, Nemeth B, Szendi K, Varga C. Clinical improvement of patients with osteoarthritis using thermal mineral water at Szigetvar Spa-results of a randomised double-blind controlled study. Int J Biometeorol. 2018 Feb;62(2):253-259. doi: 10.1007/s00484-017-1446-6. Epub 2017 Sep 27. PMID 28956169
- [Background] Hanzel A, Berenyi K, Horvath K, Szendi K, Nemeth B, Varga C. Evidence for the therapeutic effect of the organic content in Szigetvar thermal water on osteoarthritis: a double-blind, randomized, controlled clinical trial. Int J Biometeorol. 2019 Apr;63(4):449-458. doi: 10.1007/s00484-019-01676-3. Epub 2019 Feb 7. PMID 30734126